CLINICAL TRIAL: NCT02354716
Title: Expanding the Clinical Applications of Functional Luminal Imaging (EndoFLIP) in Esophageal Stenoses
Brief Title: EndoFLIP Use in Upper GI Tract Stenosis
Acronym: EndoFLIP
Status: Terminated | Type: Observational
Why Stopped: Lack of patient population
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 819014
Record Dates: First submitted 2014-12-08; First posted 2015-02-03 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Esophageal Stricture; Eosinophilic Esophagitis; Zenkers Diverticulum; Schatzki Ring
Keywords: esophagus; upper GI; endoscopy; endoFLIP; functional luminal imaging; esophageal stricture; narrow esophagus; narrow caliber esophagus; esophageal narrowing; eosinophilic esophagitis; Zenkers diverticulum; Schatzki ring
MeSH Terms: conditions — Esophageal Stenosis; Eosinophilic Esophagitis; Zenker Diverticulum

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EndoFLIP Measurements: To define the role of a functional luminal imaging probe (EndoFLIP) in benign upper GI luminal narrowing. EndoFlip measurement of the cross sectional area of the narrowing will be obtained prior to and after endoscopic dilation. Patients will follow up for repeat endoscopy and dilation if indicated. EndoFLIP measurements will be made again before and after dilation. The use of EndoFlip may offer insight in to the clinical and endoscopic predictors of successful stricture dilation.
  Interventions: Device: EndoFLIP

INTERVENTIONS:
Device: EndoFLIP — The Endolumenal Functional Lumenal Imaging Probe Imaging System is a technology developed to measure the dimensions & function of a variety of hollow organs throughout the body. Since receiving FDA clearance for sale in the United States EndoFLIP has been used in a variety of clinical applications. We intend to investigate the potential clinical applications of EndoFLIP in the upper GI tract in patients with esophageal stenoses who require endoscopic therapy for benign esophageal strictures. The use of EndoFLIP to characterize a stricture pre- & post- dilation may offer insight in to the clinical and endoscopic predictors of successful stricture dilation, & what characteristics determine & predict refractory & recurrent strictures.
  Other Names: Endolumenal Functional Lumenal Imaging Probe

SUMMARY:
The purpose of this study is to investigate the use of a functional luminal imaging probe to characterize benign esophageal luminal strictures before and after dilation and identify predictors of response to therapy. Patients will be evaluated during endoscopy using functional luminal imaging (EndoFLIP; Crospon Medical Devices, Galway, Ireland) to characterize the geometry of benign luminal esophageal narrowing before and after dilation.

DETAILED DESCRIPTION:
To date there is no effective way to objectively characterize and predict response to endoscopic dilation of luminal strictures of the GI tract. Endoscopic dilation allows effective remediation of benign esophageal and upper GI tract strictures. Stricture dilation is performed after the stricture diameter is crudely gauged by the endoscopist. Stricture characteristics are based on the severity of symptoms and appearance. A stricture may be graded as mild, moderate, severe and as to whether or not the endoscope is able to traverse the luminal narrowing. By precisely measuring the diameter and length of a stricture, the endoscopist can know exactly what type of dilation is necessary. Benign esophageal strictures may also be refractory to dilation and thus require multiple sessions, prior to achieving successful remediation. The purpose of this study is to investigate the use of a functional luminal imaging probe to characterize benign esophageal luminal strictures before and after dilation and identify predictors of response to therapy. Patients will be evaluated during endoscopy using functional luminal imaging (EndoFLIP; Crospon Medical Devices, Galway, Ireland) to characterize the geometry of benign luminal esophageal narrowing before and after dilation. The study will include patients with strictures referred for endoscopic dilation for the following indications: radiation induced strictures, peptic strictures, RFA induced strictures, EMR induced strictures, eosinophilic esophagitis, Zenkers diverticulum, and strictures related to surgical anastomoses. In patients with benign refractory esophageal strictures referred for endoluminal prostheses EndoFLIP will be used to characterize the stricture prior to stent placement.

ELIGIBILITY:
Inclusion Criteria:

* > or = to 18 years of age
* Referred for evaluation and treatment of benign esophageal luminal narrowing
* Clinical diagnosis of benign esophageal luminal narrowing with documentation and imaging
* Adult patients with benign refractory esophageal strictures referred for placement of an esophageal stent are eligible for this study
* Willing and able to give informed consent
* No condition or comorbidity which would prevent the patient from undergoing a successful upper endoscopy

Exclusion Criteria:

* < 18 years of age
* Pregnancy
* History of prior endoscopic dilation* (*unless referred for placement of stent)
* Coagulopathy
* Inability to traverse the stricture using standard techniques
* Patients unable to provide consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with benign refractory esophageal strictures referred for placement of an esophageal stent are eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Collection of Measurements of the Luminal Narrowing Using EndoFlip | 12 Months
  The study is observational and a proof of concept study. Measurements of the luminal narrowing using EndoFLIP will be obtained.

SECONDARY OUTCOMES:
Observation of Pre-Endoscopic Therapy EndoFLIP Measurements | 12 Months
  Patients will undergo the clinically indicated procedure for benign esophageal luminal narrowing remediation. Before undergoing clinically indicated esophageal therapy, measurements of the luminal narrowing using EndoFLIP will be obtained to identify potential predictors of response to endoscopic therapy. These measurements will included luminal diameter, length of narrowing and narrowing distensibility and will be obtained before and after delivery of the clinically indicated endoscopic therapy.
Observation of Post-Endoscopic Therapy EndoFLIP Measurements | 12 Months
  After undergoing clinically indicated esophageal therapy at clinically-indicated follow-up endoscopies, measurements of the luminal narrowing using EndoFLIP will again be obtained to identify responses to endoscopic therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Kochman, MD, Principal Investigator — University of Pennsylvania; Vinay Chandrasekhara, MD, Principal Investigator — University of Pennsylvania; Gregory G Ginsberg, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States